CLINICAL TRIAL: NCT00060294
Title: Phase I Study of Zevalin (90Y-Ibritumomab Tiuxetan) in Waldenstrom's Macroglobulinemia (Lymphoplasmacytic Lymphoma)
Brief Title: Yttrium Y 90 Ibritumomab Tiuxetan in Treating Patients With Waldenstrom's Macroglobulinemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: no accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000301591; UCLA-0202063; IDEC-UCLA-0202063
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Lymphoma
Keywords: Waldenström macroglobulinemia
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia | interventions — Rituximab; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: rituximab
Radiation: yttrium Y 90 ibritumomab tiuxetan

SUMMARY:
RATIONALE: Monoclonal antibodies such as yttrium Y 90 ibritumomab tiuxetan and rituximab can locate cancer cells and either kill them or deliver radioactive cancer-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of yttrium Y 90 ibritumomab tiuxetan in treating patients who have Waldenstrom's macroglobulinemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of yttrium Y 90 ibritumomab tiuxetan in patients with Waldenstrom's macroglobulinemia.
* Determine, preliminarily, the response of patients treated with this drug.

OUTLINE: This is a multicenter, dose-escalation study of yttrium Y 90 ibritumomab tiuxetan (IDEC-Y2B8).

Patients receive rituximab IV and indium In 111 ibritumomab tiuxetan (IDEC-In2B8) IV over 10 minutes on day 1. Patients then undergo gamma camera scans within 2-24 hours. Approximately 7-14 days after IDEC-In2B8, patients receive rituximab IV and IDEC-Y2B8 IV over 10 minutes. Treatment with IDEC-Y2B8 may repeat every 12 weeks in the absence of unacceptable toxicity or the achievement of a maximum cumulative dose.

Cohorts of 3-6 patients receive escalating doses of IDEC-Y2B8 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 4 years.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Waldenstrom's macroglobulinemia confirmed by IgM gammopathy and bone marrow biopsy

  * Presence of lymphoplasmacytic cells
  * CD20+ plasma cell dyscrasia on the majority of malignant cells
  * Bone marrow involvement of 20-50% by core needle biopsy of at least 1.5 cm in length
* Clinical indication for initiation of treatment, including 1 or more of the following characteristics:

  * Symptoms associated with the disease (e.g., fatigue, asthenia, or painful adenopathy)
  * Anemia
  * IgM greater than 3 g/L
  * Progression as indicated by a rate of IgM rise of more than 0.5 g over 6 months
* No myelodysplastic syndromes or profound hypocellularity of the bone marrow

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* WHO 0-2

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count greater than 1,500/mm^3
* Total B-lymphocyte count less than 5,000/mm^3
* Platelet count greater than 100,000/mm^3
* No hyperviscosity syndrome

Hepatic

* Bilirubin no greater than 1.5 mg/dL

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 year after study completion
* No uncontrolled CNS disease
* No serious nonmalignant disease that would preclude study participation
* No other concurrent active malignancy except controlled skin cancer or prostate cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 2 weeks since prior filgrastim (G-CSF) or sargramostim (GM-CSF)
* More than 4 months since prior rituximab
* No prior radioimmunotherapy

Chemotherapy

* No prior high-dose chemotherapy (unless patient has had prior back-up stem cell collections)
* More than 6 weeks since prior chemotherapy

Endocrine therapy

* More than 4 weeks since prior corticosteroids

Radiotherapy

* No prior radiotherapy

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-04; Primary Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos E. Emmanouilides, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts